CLINICAL TRIAL: NCT05127499
Title: The Effect of Progressive Relaxation Exercises Applied to Patients With Epilepsy on Depression, Sleep and Quality of Life
Brief Title: The Effect of Progressive Relaxation Exercises Applied to Patients With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Ataturk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-97132852-050.01.04-87886
Record Dates: First submitted 2021-11-03; First posted 2021-11-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; depression; progressive relaxation exercises; sleep quality of life
MeSH Terms: conditions — Epilepsy; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): will do progressive relaxation exercises
  Interventions: Other: progressive relaxation exercises
- No Intervention (No Intervention): won't do progressive relaxation exercises

INTERVENTIONS:
Other: progressive relaxation exercises — progressive relaxation exercises will do
  Arms: Experimental:

SUMMARY:
Epilepsy; It is a disease characterized by sudden, repetitive, epileptic seizures that are not triggered by an identifiable event and occur as a result of abnormal and excessive electrical discharge in cortical neurons from ancient times to the present. It is known that epilepsy has important social and psychological effects. Seizure recurrence and fear of social exclusion are life-threatening factors for epilepsy patients. These difficulties negatively affect the quality of life of patients by causing high levels of anxiety, depression, sleep disorders and low self-esteem. Many positive effects of progressive relaxation exercises on anxiety, depression, sleep and quality of life have been observed. The aim of this study is to examine the effects of progressive relaxation exercises applied to epilepsy patients on depression, sleep and quality of life.

This study, which was planned as an experimental study with a pretest-posttest control group, will be carried out by randomly dividing 60 patients diagnosed with epilepsy, who applied to the Neurology Outpatient Clinic and Clinic of Fırat University Hospital, between September 2021 and June 2022, into 2 groups as intervention and control groups. Written consent will be obtained from the patients who agreed to participate in the study at the beginning of the study, and the study will begin. Before any intervention is made in the intervention group and control group, a pre-test will be performed using the Patient Information Form, Beck Depression Scale, Pitssburg Sleep Quality Index, and Quality of Life Scale (QOLIE 31) to evaluate depression, sleep and quality of life of these patients. The intervention group will be given progressive relaxation exercises 3 times a week for 4 weeks and the control group will not make any interventions. With the posttest, both the intervention and control groups will be filled with the Patient Information FormBeck Depression Scale, Pitssburg Sleep Quality and Quality of Life Scale (QOLIE 31) and depression, sleep and quality of life will be evaluated. Finally, it will be checked whether there is a significant difference between the pretest and the posttest.

DETAILED DESCRIPTION:
epilepsy ; It is a condition characterized by sudden, repetitive, epileptic seizures that are not triggered by an identifiable event, resulting from abnormal and excessive electrical discharge in cortical neurons from ancient times to the present. In other words, epilepsy is one of the most common and chronic serious neurological diseases that require significant behavioral and psychosocial adjustments, for which a high quality of life is aimed by keeping seizures under control. In the study conducted by Rousseau et al. on 8 epileptic subjects, it was observed that the progressive relaxation exercises they applied decreased the frequency of seizures and increased the sense of well-being. It was found that it caused significant decreases in the level of depression. There is no study in the literature examining the Effect of Progressive Relaxation Exercises Applied to Epilepsy Patients on Depression, Sleep and Quality of Life. For this reason, it was aimed to examine the effects of progressive relaxation exercises applied to epilepsy patients on depression, sleep and quality of life by conducting an experimental study with a pretest-posttest control group.

ELIGIBILITY:
Inclusion Criteria:

* 55 ≤age ≥18
* Ability to communicate adequately
* Not having a diagnosed psychiatric disorder,
* Those who are determined by the physician that they do not have a physical disability in exercising
* Volunteering to participate in the research
* Individuals who have the ability to use technological tools
* A score of >5 on the Pittsburgh Sleep Quality Scale
* Having a score of >9 on the Beck Depression Scale

Exclusion Criteria:

* Those who have communication problems
* Those with psychiatric problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 4 week
  Pitssburg Sleep Quality Index, Buysse et al. It is a scale that gives a quantitative measure of sleep quality for the purpose of defining good and bad sleep. It includes a total of 24 questions. 19 of these questions are self-evaluation questions, five of which are answered by the spouse or a roommate. When calculating the index score, questions answered by the individual's spouse or roommate are not included in the calculation.The scale total score clearly distinguishes good sleepers (Scale total score ≤5) from poor sleepers (Scale >5)
Beck Depression Scale | 4 week
  It is a self-assessment type scale developed by Beck et al. (1961) to measure the level of depression symptoms and change in severity in the adult age group. The Turkish validity and reliability study was performed by Hisli (1988). It consists of 21 items that measure the symptoms in the vegetative, emotional, cognitive and motivational areas of depression.Minimal depression 0-9, Mild depression 10-16, Moderate depression 17-29, Severe depression 30-63
Quality of Life in Epilepsy-31 | 4 week
  Its validity and reliability have been verified by Mollaoğlu et al.. Only epilepsy-related issues are questioned in the scale. It consists of 7 sub-dimensions. These sub-dimensions are; seizure anxiety (5 items), emotional well-being (5 items), energy/fatigue (4 items), social function (5 items), cognitive function (6 items), effects of drugs (3 items), total quality of life (2 items) and an additional item evaluating the total health status. The scale is scored between 0-100. A high score reflects a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahcecioglu Turan, PhD, Study Chair — Firat University
Locations (1):
- Fırat Üniversitesi, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Controlled Examination of Effects of Progressive Relaxation Training on Seizure Reduction — https://pubmed.ncbi.nlm.nih.gov/1628583/